CLINICAL TRIAL: NCT03878238
Title: Randomized, Double Blind and Placebo-controlled Pilot Study to Evaluate the Effect of a Probiotic Mixture in Acne Vulgaris
Brief Title: A Pilot Study to Evaluate the Effect of a Probiotic Mixture in Acne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bionou Research, S.L. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACNE_PROB
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Acne; Acne Vulgaris
Keywords: Probiotic
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Probiotic (Experimental)
  Interventions: Dietary Supplement: Probiotic Bths-003

INTERVENTIONS:
Dietary Supplement: Probiotic Bths-003 — Probiotic with maltodextrin as a carrier.
  Arms: Probiotic
Other: Placebo — Placebo with maltodextrin base.
  Arms: Placebo

SUMMARY:
A 12-week randomized, double-blind, placebo-controlled pilot study to evaluate the effect of a probiotic blend in the treatment and clinical and subjective evolution of acne vulgaris in adolescent and adult patients between 12 and 30 years.

ELIGIBILITY:
Inclusion Criteria:

* Signature of informed consent by the patient (and their legal guardian in case of being under age).
* Age between 12 and 30 years-old.
* Moderate acne according to the AGSS (Acne Global Severity Scale) and / or GAGS (Global Acne Grading System) scales.

Exclusion Criteria:

* Contraindication of any of the components of the product under study.
* Topical or systemic use of antifungals and antibiotics in the previous 2 weeks.
* Consumption of probiotics in the previous 2 months.
* Use of systemic retinoids in the previous 6 months.

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-05-29 (Actual)

PRIMARY OUTCOMES:
Change from baseline in GAGS (Global Acne Grading System) index score at 12 weeks | 12-week
  TOTAL SCORE = Nose S x 1 + Chin S x 1 + Front S x 2 + Right cheek S x 2 + Left cheek S x 2 + Torso S x 3
  [Severity (S): 0 = Absence; 1 = Comedones; 2 = Papules; 3 = Pustules; 4 = Nodules]
  SCORE: 0 = Clean; 1-18 = Mild; 19-30 = Moderate; 31-38 = Severe; > 38 = Very severe

SECONDARY OUTCOMES:
AGSS (Acne Global Severity Scale) index score | 0, 6 and 12-week
  Score between 0 and 5:
  0 = Clean = Normal and clear skin without evidence of acne
  1. = Almost clean = There are some non-inflammatory lesions, with uncommon and non-inflamed papules
  2. = Mild = few inflammatory lesions (no nodule-cystic lesions)
  3. = Moderate = Noninflammatory lesions predominate, but multiple inflammatory lesions appear (nodule-cystic lesions may be present)
  4. = Severe = Inflammatory lesions predominate (nodule-cystic lesions may be present)
  5. = Very severe = Highly inflammatory lesions predominate (several nodule-cystic lesions)
Number of acne lesions | 0, 6 and 12-week
  Number of non-inflammatory, inflammatory and total acne lesions.
Patient subjective evaluation | 0, 6 and 12-week
  Min score (Best) = 6 Max score (Worst) = 30
Adherence to treatment | 12-week
  Compliance rate (in percentage) calculated as the number of leftover capsules divided by the total number of days between visits.
Treatment safety assessed by number of adverse events | 12-week
  Number of adverse events that occur during the treatment period.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Vithas Nisa 9 de Octubre, Valencia, Spain